CLINICAL TRIAL: NCT03846960
Title: Surfactant Administration Via Thin Catheter Using a Specially Adapted Video Laryngoscope - a Prospective Study Assessing the Feasibility of the VISUAL (Video Surfactant Administration Laryngoscopy) Method
Brief Title: Surfactant Administration Via Thin Catheter Using a Specially Adapted Video Laryngoscope
Acronym: VISUAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Gil Talmon, Senior Attending Neonatologist, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0149-18-EMC
Record Dates: First submitted 2019-01-08; First posted 2019-02-20 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Distress Syndrome
Keywords: video laryngoscope; minimally invasive surfactant administration
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Thiosulfate Sulfurtransferase

STUDY DESIGN:
Intervention Model Description: intervention of a device product being evaluated in a small clinical trial to determine the feasibility of the product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- preterm infants (Experimental): A prospective study to assess the safety and efficacy of surfactant administration via thin catheter using a specially adapted VNscope, originally used for endotracheal intubation and adapted for the administration of surfactant without the placement of an endotracheal tube. A feasibility study of 10 preterm infants 30-36 gestational age at birth, that requires surfactant administration for the indication of respiratory distress syndrome, and do not require immediate intubation
  Interventions: Device: using specially adapted VNscope; Drug: surfactant administration

INTERVENTIONS:
Device: using specially adapted VNscope — surfactant administration via thin catheter using a specially adapted VNscope
  Other Names: VNScope VNS0-000; VNBlade VNB0-000/1
Drug: surfactant administration — surfactant administration via thin catheter using a specially adapted VNscope
  Other Names: Curosurf - a porcine surfactant routinely used for RDS

SUMMARY:
In this study the investigators intend to assess the feasibility of surfactant administration via a thin catheter using a specially adapted video laryngoscope, with a groove designed to allow insertion of an endovascular catheter without the use of other instruments in the oral cavity (forceps ect.). The laryngoscope is of Peak Medic Ltd, Netania, Israel.

DETAILED DESCRIPTION:
A prospective study to assess the safety and efficacy of surfactant administration via thin catheter using a specially adapted VNscope, originally used for endotracheal intubation and adapted for the administration of surfactant without the placement of an endotracheal tube.

Once neonates present respiratory distress, the adapted scope will be used - clinical and outcome measures will be collected to asses the safety and efficacy of the use

ELIGIBILITY:
Inclusion Criteria:

1. - Premature infants with gestational age 30-36 weeks.
2. - Diagnosis of respiratory distress syndrome
3. - Treatment with antenatal steroids.
4. - Spontaneously breathing with non-invasive positive pressure ventilation.
5. - maximal age 3 days.

Exclusion Criteria:

1. - Apgar score at 5 min < 5
2. - Need for chest compressions or medication upon delivery.
3. - Evident major congenital malformation, metabolic or genetic disorders.
4. - Clinical evidence of sepsis.

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of attempts until surfactant is administrated | maximal age 3 days.
  Number of intubation attempts- higher values represent a worse outcome
Assessment of the infants' stability during the procedure - saturation, bradycardia, tachycardia. | maximal age 3 days.
  Monitoring the baby during the procedure and assessment of the infants' stability:
  hypoxia (Oxygen saturation less than 60% for more than 5 sec), bradycardia (HR less than 60 for more than 5 sec), tachycardia (HR more than 220 for more than 5 sec) bradycardia below 100 bpm and tachycardia above 220 bpm indicate worse outcome
Duration of the entire procedure, form laryngoscope insertion to surfactants administration and Laryngoscope blade out of the mouth. | maximal age 3 days.
  Time measurement of the procedure, sorter time indicate a better outcome

SECONDARY OUTCOMES:
Need of invasive mechanical ventilation in the next 24 hours. | maximal age 3 days.
  Failure of non-invasive approach and conversion to invasive ventilation to evaluate the efficiency of the procedure
complications reports - one lung surfactant administration, pneumothorax, NEC, IVH, Pulmonary Hemorrhage | maximal age 3 days.
  Documentation of the complication related to the procedure according to the clinical signs and chest x-ray after the procedure
Subjective procedure scale of assessment. | maximal age 3 days.
  Physician subjective assessment to evaluate the feasibility of the procedure- IRB- approved survey aims to assess user experiences with Video Surfactant Administration Laryngoscopy method in NICU. The survey contains five levels- a) Very satisfied b) Somewhat satisfied c) Neither satisfied nor dissatisfied d) Somewhat dissatisfied e) Very dissatisfied
Unexpected pitfalls reports | maximal age 3 days.
  Physician assessment to evaluate eny pitfalls during the procedure
Safety assessment of the procedure (Physician questionnaire) | maximal age 3 days.
  Physician questionnaire- Do you feel VISUAL method is safe for the premature baby?
  a)Yes b)Maybe c)No

CONTACTS AND LOCATIONS:
Overall Officials: Gil talmon, dr, Principal Investigator — haemek medical center
Locations (1):
- Haemek medical centre, Afula, Israel